CLINICAL TRIAL: NCT04561583
Title: A Prospective, Multi-center, Single-blind, Parallel, Randomized Controlled Clinical Trial Designed to Evaluate the Safety and Effectiveness of the LED Light Source System for Endoscope During Ureter Transillumination.
Brief Title: Effectiveness and Safety of LED Light Source System for Endoscope
Acronym: ENV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was registered but never started.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Stryker02
Record Dates: First submitted 2020-09-01; First posted 2020-09-23 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: gallstone; cholecystitis; gallbladder polyp
MeSH Terms: conditions — Gallstones; Cholecystitis | interventions — Endoscopes

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, multi-center, single-blind, parallel, randomized controlled clinical trial. The trial will be carried out in 5 centers, involving 220 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 110 subjects).
  This trial will be carried out in 4 stages, including the screening period, random grouping, operation date and follow-up period. In the screening period, the informed consent forms are collected and inclusion and exclusion criteria are verified; after that, the accepted subjects will be randomly divided into the control group or test group; on the operation date, the operation is carried out using the device; safety follow-up visit is carried out during the follow-up period.
Who Masked: Participant
Masking Description: In this trial, single-blind method will be used, which means that the investigators know about the device used for treatment of the subjects while the subjects know nothing about it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LED light source system for endoscope (Other): This trial is designed as a prospective, multi-center, single-blind, parallel, randomized controlled clinical trial. The trial will be carried out in 5 centers, involving 220 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 110 subjects).Test grop use LED light source system for endoscope
  Interventions: Device: LED light source system for endoscope
- Pinpoint Endoscopic Fluorescence Imaging System (Other): This trial is designed as a prospective, multi-center, single-blind, parallel, randomized controlled clinical trial. The trial will be carried out in 5 centers, involving 220 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 110 subjects).control group use Pinpoint Endoscopic Fluorescence Imaging System (Model: PC9000)
  Interventions: Device: Pinpoint Endoscopic Fluorescence Imaging System

INTERVENTIONS:
Device: LED light source system for endoscope — This trial is designed as a prospective, multi-center, single-blind, parallel, randomized controlled clinical trial. The trial will be carried out in 5 centers, involving 220 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 110 subjects).
  This trial will be carried out in 4 stages, including the screening period, random grouping, operation date and follow-up period. In the screening period, the informed consent forms are collected and inclusion and exclusion criteria are verified; after that, the accepted subjects will be randomly divided into the control group or test group; on the operation date, the operation is carried out using the device; safety follow-up visit is carried out during the follow-up period.
  Arms: LED light source system for endoscope
Device: Pinpoint Endoscopic Fluorescence Imaging System — This trial is designed as a prospective, multi-center, single-blind, parallel, randomized controlled clinical trial. The trial will be carried out in 5 centers, involving 220 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 110 subjects).
  This trial will be carried out in 4 stages, including the screening period, random grouping, operation date and follow-up period. In the screening period, the informed consent forms are collected and inclusion and exclusion criteria are verified; after that, the accepted subjects will be randomly divided into the control group or test group; on the operation date, the operation is carried out using the device; safety follow-up visit is carried out during the follow-up period.
  Arms: Pinpoint Endoscopic Fluorescence Imaging System

SUMMARY:
This trial is designed as a prospective, multi-center, single-blind, parallel, randomized controlled clinical trial. The trial will be carried out in 5 centers, involving 220 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 110 subjects).

This trial will be carried out in 4 stages, including the screening period, random grouping, operation date and follow-up period. In the screening period, the informed consent forms are collected and inclusion and exclusion criteria are verified; after that, the accepted subjects will be randomly divided into the control group or test group; on the operation date, the operation is carried out using the device; safety follow-up visit is carried out during the follow-up period.

DETAILED DESCRIPTION:
The prospective, multi-center, single-blind, parallel, randomized controlled non-inferiority trial design is adopted to evaluate the safety and effectiveness of the real-time endoscopic near infrared fluorescence image provided by the LED light source system for endoscope by evaluating at least one main extrahepatic bile duct (common bile duct and ductuli hepaticus communis). The trial will be carried out in 5 centers, with the competitive grouping mode adopted. Totally 220 patients to receive laparoscopic cholecystectomy will be involved (110 patients for each of the control group and the test group). The subjects, after signing the informed consent form approved by the Ethics Committee, will be screened by the investigators. Qualified subjects who meet all the inclusion criteria and do not meet any of the exclusion criteria will be randomly divided into the control group or the test group. For the subjects in the control group, the Pinpoint Endoscopic Fluorescence Imaging System commercially available will be used for operation. For subjects of the test group, the LED light source system for endoscope will be used for operation. On the operation date, investigators will evaluate the display performance of the device by judging whether at least one main extrahepatic bile duct (common bile duct and ductuli hepaticus communis) is displayed. During the follow-up period, the investigators will evaluate the safety of the device based on the results of vital signs, physical examination, blood routine examination, routine urine examination, blood biochemistry and 12-lead ECG.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Subjects who should receive laparoscopic cholecystectomy on a selected day Symptoms of such subjects include gallstone, cholecystitis, or gallbladder polyp≥0.8 cm
   2. Aged between 18 and 75
   3. All subjects voluntarily participate in the clinical trial and are asked to sign the informed consent form
2. Exclusion Criteria:

   1. Subjects suffering acute cholecystitis and cholangitis
   2. Subjects requiring laparotomy
   3. Women during pregnancy or lactation
   4. Subjects expected to give birth to a child within 3 months after the trial
   5. Subjects suffering liver cirrhosis
   6. Subjects allergic to ICG or iodine
   7. Subjects with cardiopulmonary insufficiency and those intolerant of surgery
   8. Subjects with abnormal renal and liver function: ①Aspartate aminotransferase AST or alanine aminotransferase ALT exceeding 3 times of the upper limit of the normal range; ② Serum creatinine > 2.0 mg/dL or ≥ 176.8 μmol/L
   9. Subjects with history of malignant cancer or subjects with malignant cancer
   10. Subjects currently engaged in other clinical trials
   11. Subjects deemed by the investigators as unsuitable for the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Visualization rate of extrahepatic bile duct. | During the operation
  Note: The visualization rate of extrahepatic bile duct refers to the visualization rate of at least one extrahepatic bile duct (the ductuli hepaticus communis and common bile duct) after dissection of the calot's triangle (the images are taken respectively before unfolding the anatomical structure, during dissection and after complete unfolding of the triangular structure).

SECONDARY OUTCOMES:
Time of operation | During the operation
  Time of operation
Intraoperative blood loss | During the operation
  Intraoperative blood loss
the occurrence rate of complications | Postoperative follow-up period was up to 7 days
  bile duct injury, bile leakage, hemorrhage, secondary abdominal infection
Device failure rate | During the operation
  Device failure rate

OTHER OUTCOMES:
adverse events | Informed to sign into the interview window 7 days after surgery
  Incidence (%) and frequency (number of events) of adverse events
serious adverse events | Informed to sign into the interview window 7 days after surgery
  Incidence (%) and frequency (number of events) of serious adverse events
device-related adverse events | Informed to sign into the interview window 7 days after surgery
  Incidence (%) and frequency (number of events) of device-related adverse events
serious device-related adverse events | Informed to sign into the interview window 7 days after surgery
  Incidence (%) and frequency (number of events) of serious device-related adverse events
device deficiency | During the operation
  Incidence (%) and frequency (number of events) of device deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (4):
- China (4):
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol will be shared
Supporting Information: Study Protocol
Time Frame: The clinical trial begins and ends
Access Criteria: From the beginning to the end of the clinical trial, the participating centers followed the protocol of consent